CLINICAL TRIAL: NCT06605118
Title: Azithromycin Prophylaxis for Prelabor Cesarean Delivery Trial
Acronym: PRECEDE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD036801-PRECEDE; U01HD114634 (NIH); U24HD036801 (NIH)
Record Dates: First submitted 2024-09-13; First posted 2024-09-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Obstetrical Complications; Labor and Delivery Complication; Cesarean Delivery
Keywords: cesarean delivery; infection; maternal morbidity; antibiotics; prevention
MeSH Terms: conditions — Infections | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized shortly before delivery to receive either azithromycin administered intravenously or a placebo control of normal saline administered intravenously
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study medication will be prepared by the center research pharmacies from a list provided by the independent data coordinating center, with the active and placebo medication having identical appearance. No other individuals, including the participant or any other clinical or research staff will be informed of the study assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azithromycin prophylaxis and standard of care preoperative antibiotics (Experimental): 500mg of intravenous azithromycin administered up to 1 hour prior to cesarean incision (or as soon as feasible after incision) and infused over one hour per FDA infusion recommendations for azithromycin. Additionally patients will received standard of care preoperative antibiotics (excluding azithromycin) prior to incision.
  Interventions: Drug: Azithromycin Injection; Drug: Standard of Care Preoperative antibiotics
- Placebo and standard of care preoperative antibiotics (Placebo Comparator): Normal saline administered up to 1 hour prior to cesarean incision (or as soon as feasible after incision) and infused over one hour in addition to standard of care preoperative antibiotics (excluding azithromycin) prior to incision.
  Interventions: Drug: Placebo; Drug: Standard of Care Preoperative antibiotics

INTERVENTIONS:
Drug: Azithromycin Injection — 500mg azithromycin in 250 mL of normal saline
  Arms: Azithromycin prophylaxis and standard of care preoperative antibiotics
Drug: Placebo — 250 mL of normal saline
  Arms: Placebo and standard of care preoperative antibiotics
Drug: Standard of Care Preoperative antibiotics — standard of care preoperative antibiotics (excluding azithromycin) prior to incision

SUMMARY:
This is a phase-III multi-center double-blind randomized controlled trial of 8,000 individuals undergoing a scheduled or prelabor cesarean delivery who are randomized to either adjunctive azithromycin prophylaxis or to placebo. Both groups also will receive standard of care preoperative antibiotics (excluding azithromycin). The primary endpoint is a maternal infection composite defined as any one of the following up to 6 weeks postpartum: endometritis, wound infection, abscess, septic thrombosis, sepsis, pneumonia, pyelonephritis and breast infection.

DETAILED DESCRIPTION:
This is a phase-III multi-center double-blind randomized controlled trial of 8,000 individuals undergoing a scheduled or prelabor cesarean delivery who are randomized to either azithromycin prophylaxis or to placebo. All participants will receive standard of care preoperative antibiotics. The primary objective is to evaluate in patients undergoing scheduled/prelabor cesarean if pre-incision adjunctive azithromycin prophylaxis reduces the risk of post-cesarean infections compared with placebo. Secondary objectives include 1) to assess the perinatal and maternal safety of pre-incision adjunctive azithromycin, 2) to evaluate whether adjunctive azithromycin prophylaxis reduces maternal and neonatal resource use outcomes compared with placebo, and 3) to evaluate whether adjunctive azithromycin influences maternal and neonatal infection with resistant organisms compared with placebo.

Individuals will be randomized prior to the start of the cesarean to either 500mg of intravenous azithromycin or to placebo (normal saline). Maternal blood and cord blood will be collected on a subset of the population. Research staff will abstract maternal and neonatal outcomes following delivery and discharge from the hospital. A single maternal follow-up study visit at 6 weeks (4-8 weeks) postpartum will be scheduled to ascertain maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 23 weeks' gestation (ACOG dating criteria)
* Scheduled or prelabor cesarean delivery
* Singleton or twin gestation

Exclusion Criteria:

* Allergy or contraindication to azithromycin or macrolide antibiotics, including those with a history of cholestatic jaundice/hepatic dysfunction associated with prior use of azithromycin
* Chorioamnionitis
* Bacterial infection (e.g., pyelonephritis) requiring ongoing antibiotic treatment after delivery
* Premature rupture of membranes (PROM) or labor (i.e., contractions with ongoing cervical change)
* Fetal demise or known major congenital anomaly
* Azithromycin treatment within 7 days
* Planned use of antimicrobial prophylaxis after delivery for any reason
* Known structural heart disease or active cardiomyopathy (current ejection fraction<40%)
* Known arrhythmia with QT prolongation or taking scheduled medications known to prolong the QT interval such that it would preclude the use of azithromycin
* Refusal or unable to obtain consent (e.g., language barrier)
* Participating in another intervention study that influences the primary outcome in this study
* Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, do not have to be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Maternal infection composite | Delivery up to 6 weeks postpartum (a period of up to 6 weeks)
  a maternal infection composite defined as any one of the following: endometritis, wound infection, abdominal or pelvic abscess, septic pelvic thrombosis, sepsis, pneumonia, pyelonephritis and breast infection

SECONDARY OUTCOMES:
Non-infections wound complications | Delivery up to 6 weeks postpartum (a period of up to 6 weeks)
  any of the following wound complications without diagnosis of a wound infection: seroma, wound breakdown, erythema and/or hematoma
Perinatal composite outcome | hospital discharge, 6 weeks of birth, or death (whichever occurs first)
  Any of the following:
  * Neonatal death occurring within 28 days of birth or prior to initial discharge from hospital
  * Respiratory distress syndrome
  * Necrotizing enterocolitis grade 2 or higher
  * Periventricular leucomalacia
  * Intraventricular hemorrhage grades 3 or 4
  * Bronchopulmonary dysplasia grade 3 or higher
  * Suspected sepsis
  * Confirmed sepsis
  * Cardiac resuscitation
  * Severe neonatal drug reaction defined as anaphylaxis or any other reported severe event suspected to be due to azithromycin
  * Hypertrophic pyloric stenosis defined as physician diagnosis supported by surgical intervention (pyloromyotomy) or pathology evaluation through 6 weeks from birth.
Number of neonates with Allergic Reaction | birth through hospital discharge, or 7 days from birth, whichever is earliest
  Neonatal allergic reaction (e.g., skin rash) through discharge or 7 days from birth, whichever is earliest, suspected to be due to study medication.
Number of Neonates with Gastrointestinal Symptoms | birth through hospital discharge, or 7 days from birth, whichever is earliest
  vomiting, diarrhea, feeding difficulty through discharge or 7 days from birth, whichever is earliest
Number of Maternal Deaths | From randomization through 6 weeks postpartum (a period of up to 6 weeks)
  Death
Maternal Resource Composite | From hospital discharge following delivery through 6 weeks postpartum (a period of up to 6 weeks)
  * Hospital readmission
  * Emergency room (ER) visit
  * Unscheduled clinic visits
Neonatal Resource Composite | From hospital discharge following delivery through 6 weeks postpartum (a period of up to 6 weeks)
  * Hospital readmission
  * Emergency Room (ER) visit
Maternal Hospital Length of Stay | Hospital admission to hospital discharge (up to 42 days)
  Length of hospital stay in days
Rate of Neonatal ICU Admission | Delivery to hospital discharge (up to 120 days)
  Number of neonates admitted to NICU
Number of Participants with Maternal Resistant Infection | Randomization through 6 weeks postpartum (a period of up to 6 weeks)
  bacteria and resistance patterns from clinical cultures
Number of Neonates with Neonatal Resistant Infection | From birth up to 6 weeks of age
  bacteria and resistance patterns from clinical cultures

CONTACTS AND LOCATIONS:
Overall Officials: Alan T.N. Tita, MD PhD, Study Chair — University of Alabama at Birmingham; Kim Boggess, MD, Study Chair — University of North Carolina, Chapel Hill; Monica Longo, MD PhD, Study Director — Eunice Kennedy Shriver NICHD; Rebecca G Clifton, PhD, Principal Investigator — The George Washington University Biostatistics Center
Locations (14):
- United States (14):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Regents of the University of California San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Brown Univeristy, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via NICHD DASH in accordance with NIH policy.
Supporting Information: Study Protocol, ICF